CLINICAL TRIAL: NCT01931020
Title: Double Blind Randomised Controlled Trial to Compare the Efficacy of Oral 25% Glucose With Oral 24% Sucrose for Pain Relief During Heel Lance in Preterm Neonates
Brief Title: Analgesic Effect of Oral 25% Glucose Versus Oral 24% Sucrose for Pain Relief During Heel Lance in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Principal Investigator, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Glucose versus sucrose in pain
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Pain; Preterm; Neonates; 24% Sucrose; 25% Dextrose
MeSH Terms: conditions — Pain; Premature Birth | interventions — Sucrose; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucrose (Active Comparator): 1ml of 24%sucrose will be administered prior to heel lance
  Interventions: Drug: Sucrose
- Glucose (Experimental): 1ml of 25% glucose will be administered prior to heel lance
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Sucrose — The enrolled neonates will be administered 1ml of 24% sucrose. After 2 minutes heel lancing will be performed after cleaning the heel of neonate with a sterile spirit swab, with an auto lancet. Neonate's faces and monitor screen will be filmed in real time by using two independent video cameras during the entire procedure i.e. staring 2 minutes prior to heel lance and continue 2 minutes after the procedure. The PIPP will be assessed at 30 seconds, 1 minute and 2 minute after the procedure.
  Other Names: 24% Sucrose
  Arms: Sucrose
Drug: Glucose — The enrolled neonates will be administered 1ml of 25% gluose. After 2 minutes heel lancing will be performed after cleaning the heel of neonate with a sterile spirit swab, with an auto lancet. Neonate's faces and monitor screen will be filmed in real time by using two independent video cameras during the entire procedure i.e. staring 2 minutes prior to heel lance and continue 2 minutes after the procedure. The PIPP will be assessed at 30 seconds, 1 minute and 2 minute after the procedure.
  Other Names: 25% Glucose
  Arms: Glucose

SUMMARY:
RESEARCH HYPOTHESIS-In preterm neonates during heel lance oral 25% glucose is more efficacious in reducing pain as compared to oral 24% sucrose when assessed by PIPP(Premature infant pain profile)

DETAILED DESCRIPTION:
Pain is "an unpleasant sensory and emotional experience associated with actual or potential tissue damage". Evaluation of pain in neonates is difficult due to the subjective nature of pain and the inability of neonates to verbally express pain. Surrogate measures used to describe pain in neonates include motor responses, facial expressions, cry and changes in physiologic parameters like heart rate, blood pressure, oxygen saturation and respiratory rate. Various changes have been compiled to create various scores. Validated scores for the assessment of pain include Neonatal Facial Coding System, Neonatal Infant Pain Scale or Premature Infant Pain Profile. These reactions to pain may contribute to the development of hypoxia, hypercarbia, acidosis, ventilator asynchrony, pneumothoraces, reperfusion injury and venous congestion and subsequent late intraventricular hemorrhage (IVH) or late extension of early intraventricular hemorrhage and periventricular leukomalacia. These behavioral changes may also disrupt postnatal adaptation, parent-infant bonding and feeding schedules.

Newborn infants routinely undergo painful invasive procedures, even after uncomplicated birth. Evidence shows that neonates do feel pain and may even have increased sensitivity to pain and to its long term effects compared with older infants. Treating procedural pain has become a crucial part of neonatal care. In healthy infants, the most common painful procedures are heel lance and venipuncture. Though minimally invasive, lancing is a painful procedure that activates cortical areas in brain .Repetitive procedural pain can lead to changes in the pain sensitivity threshold therefore, adequate analgesic control is needed. Pharmacological treatments are rarely used during these procedures because of concerns about their effectiveness (topical local anesthetics or paracetamol for heel pricks) and potential adverse effects (central analgesics). Therefore, non-pharmacological interventions are valuable alternatives. Recent interventions such as sweet oral solutions (sucrose or glucose) and non-nutritive sucking have been used frequently to alleviate pain.

Use of sucrose in preterm neonates has been advocated uniformly for pain relief. However, recently few reports have raised concerns over its safety and effect on neurodevelopment. Glucose has been used in pain relief in neonates but its therapeutic efficacy in comparison to oral sucrose in direct adequately powered RCT with pain assessment tools has not been evaluated in the Indian subcontinent. The present study was planned to evaluate the efficacy of 25% glucose solution with 24% sucrose solution for analgesia during heel lance in preterm neonates.

LACUNAE IN EXISTING KNOWLEDGE Existing literature on efficacy of glucose vs. sucrose is inconclusive on superiority of either. When a Medline search was carried out it returned limited results and no results returned from the Indian subcontinent which compared the two solutions using a multidimensional pain assessment tool. There is a need for an efficacious and cheap substitute which is readily available in NICU settings and sterile. Hence, the role of 25% Glucose in neonatal pain relief and safety associated with its use needs to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at <37 weeks of gestational age
* Infants within first 48 hours of post natal life
* Infants having clinical indication for blood sampling
* Parental consent

Exclusion Criteria:

* Infants born with perinatal asphyxia, birth trauma, cardiorespiratory instability
* Infants with 5min APGAR score <7
* Infants having any syndromes, congenital anomalies or previous surgery
* Infants born to mothers known to be receiving opiates
* Infants administered muscle relaxants, sedatives & analgesics
* Infants born under general anesthesia

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Painful response | 30 seconds after heel lance
  Premature Infant Pain Profile(PIPP)

SECONDARY OUTCOMES:
Duration of Crying | Within 2 minutes following the procedure
  Duration of crying will be taken as the time between the first crying sound till total silence

OTHER OUTCOMES:
Number of Participants with Adverse Events | Within 2 minutes following the procedure
  * Choking, coughing or vomiting
  * Sustained tachycardia (HR>200) for >15 seconds
  * Sustained bradycardia (HR<80) for >15 seconds
  * Sustained tachypnea (RR>80) for >15 seconds
  * Sustained dyspnea (RR<20) for >15 seconds
  * Sustained oxygen desaturation <80% for >15 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Datta, MD, Principal Investigator — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College, New Delhi, Delhi1, India

IPD SHARING:
Plan to Share IPD: Undecided